CLINICAL TRIAL: NCT06480344
Title: Risk Factors Associated With the Occurrence of Surgical Site Infections (SSI) in Patients Operated for Acute Abdomen at Hôpital de l'Université d'Etat d'Haiti (HUEH) From January 2018 to December 2020
Brief Title: Analysis of Risk Factors for Surgical Site Infections in Patients With Acute Abdomen at Hospital of State University of Haiti
Status: Completed | Type: Observational
Sponsor: University of Haiti (Other)
Collaborators: Christopher Williams Valsaint (Unknown); Axler Jean-Paul (Unknown)
Responsible Party: Principal Investigator, Thaimye Joseph, Medical Doctor, University of Haiti
Other Study IDs: JTCVCC001
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Surgical Site Infection; Post-Op Infection
Keywords: Surgical site infection; NNIS index; Post-operative infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients who developed surgical site infection.
- Controls: Patients who did not developed surgical site infection.

SUMMARY:
The purpose of this study is to identify the risk factors associated with surgical site infection.

DETAILED DESCRIPTION:
87 patients medical records from January 2018 to December 2020 will be analyzed to detect the risk factors linked to the occurence of surgical site infection. Then the strength of their association with surgical site infection will be determined via multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients over 12 years of age.
* Admitted to the Surgery Department for acute surgical abdomen and having undergone surgery

Exclusion Criteria:

* Patients who have undergone abdominal surgery for urological or gynecological pathologies
* Files with missing information on preoperative, operative and post-operative arrangements

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants selected in our study include those who have developed an infection at the operating site (case) as well as those who have not developed it (controls) following acute abdominal surgery diagnosed in post-op room at the surgery department of The State University of Haiti, from January 2018 to December 2022.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Occurence of surgical site infection | 1 year
  Wheter or not patients developed surgical site infection

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital de l'Université d'Etat d'Haiti, Port-au-Prince, Ouest, Haiti

IPD SHARING:
Plan to Share IPD: No